CLINICAL TRIAL: NCT04493008
Title: Antibiotic Usage and Resistance - A Survey on Knowledge and Practices Among Second Year Dental Students and Patients Attending Misr International University Dental Clinics Before and After Educational Sessions
Brief Title: Antibiotic Usage and Resistance; Knowledge and Practices Before and After Educational Sessions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Misr International University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PUB 2123001
Record Dates: First submitted 2020-07-27; First posted 2020-07-30 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2020-07

CONDITIONS: Antibiotics
Keywords: Antibiotic resistance; Antibiotic uses; Knowledge about antibiotics; dental students

STUDY DESIGN:
Intervention Model Description: Single group will be assessed before and after an educational session
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MIU students and patents (Other): Educational session
  Interventions: Behavioral: Experimental: Educational session

INTERVENTIONS:
Behavioral: Experimental: Educational session — Each patient will receive educational session consisting of face-to-face interview, administration of posters, brochures and pamphlets.

SUMMARY:
The inappropriate use of antibiotics by patients not only increases the growth of resistant bacterial strains but also, may lead to adverse side effects that range from gastrointestinal disturbances to fatal anaphylactic shock. To meet the challenges faced by the spread of antibiotics resistance, different approaches have been taken worldwide. One of the approaches which are commonly proposed is to engage instructional and educational campaigns among the health care personnel and the general population about antibiotic resistance and its dangerous consequences.The present study aims at assessing the knowledge, practices of antibiotic uses and resistance before and after educational sessions among second year dental students and a group of patients attending MIU Dental Clinics.

DETAILED DESCRIPTION:
Statement of problem: Dental students' and patients' knowledge about antibiotic uses are essential for overcoming antibiotic resistance. Antibiotic resistance is considered an important global public health problem and is recognized as a major cause of the emerging problem of antimicrobial agent resistance. The inappropriate use of antibiotics by patients not only increases the growth of resistant bacterial strains but also, may lead to adverse side effects that range from gastrointestinal disturbances to fatal anaphylactic shock. To meet the challenges faced by the spread of antibiotics resistance, different approaches have been taken worldwide. One of the approaches which are commonly proposed is to engage instructional and educational campaigns among the health care personnel and the general population about antibiotic resistance and its dangerous consequences.

Aim of the study: The present study aims at assessing the knowledge, practices of antibiotic uses and resistance before and after educational sessions among second year dental students and a group of patients attending MIU Dental Clinics.

Materials and Methods: The study will be conducted on (315) second year dental students through a pre-and post-educational sessions questionnaire. Students will receive training sessions for four hours during their dental public health course given by senior staff members before conducting educational sessions targeting patients attending MIU Dental Clinics. Educational sessions will include verbal and visual tools.

ELIGIBILITY:
Inclusion Criteria:

* Second year dental students at MIU during the Academic Year 2017/2018. Any patient over 18 years old attending the MIU Dental clinics, and agreeing to sign an informed consent to participate in the study

Exclusion Criteria:

* Patients with mental disorders, deaf, and blind patients will be excluded from the study because the educational sessions will include verbal and visual tools.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Knowledge about antibiotics | 4 months
  Percentage of correct answers

SECONDARY OUTCOMES:
Awareness level | 4 months
  Percentage

CONTACTS AND LOCATIONS:
Overall Officials: Mahassen M Farghaly, Professor, Study Director — Vice president of community services and environmental awareness
Locations (1):
- Faculty of Oral & Dental Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cope AL, Wood F, Francis NA, Chestnutt IG. General dental practitioners' perceptions of antimicrobial use and resistance: a qualitative interview study. Br Dent J. 2014 Sep;217(5):E9. doi: 10.1038/sj.bdj.2014.761. PMID 25213543
- [Background] Tulip DE, Palmer NO. A retrospective investigation of the clinical management of patients attending an out of hours dental clinic in Merseyside under the new NHS dental contract. Br Dent J. 2008 Dec 20;205(12):659-64; discussion 648. doi: 10.1038/sj.bdj.2008.1044. Epub 2008 Dec 5. PMID 19057559
- [Background] Dailey YM, Martin MV. Are antibiotics being used appropriately for emergency dental treatment? Br Dent J. 2001 Oct 13;191(7):391-3. doi: 10.1038/sj.bdj.4801190. PMID 11697600
- [Background] Sweeney LC, Dave J, Chambers PA, Heritage J. Antibiotic resistance in general dental practice--a cause for concern? J Antimicrob Chemother. 2004 Apr;53(4):567-76. doi: 10.1093/jac/dkh137. Epub 2004 Feb 25. PMID 14985274
- [Background] Abu-Mostafa NA, Al-Mejlad NJ, Al-Yami AS, Al-Sakhin FZ, Al-Mudhi SA. A survey of awareness related to the use of antibiotics for dental issues among non-medical female university students in Riyadh, Saudi Arabia. J Infect Public Health. 2017 Nov-Dec;10(6):842-848. doi: 10.1016/j.jiph.2017.01.015. Epub 2017 Feb 21. PMID 28233723
- [Background] Metlay JP, Stafford RS, Singer DE. National trends in the use of antibiotics by primary care physicians for adult patients with cough. Arch Intern Med. 1998 Sep 14;158(16):1813-8. doi: 10.1001/archinte.158.16.1813. PMID 9738612
- [Background] McManus P, Hammond ML, Whicker SD, Primrose JG, Mant A, Fairall SR. Antibiotic use in the Australian community, 1990-1995. Med J Aust. 1997 Aug 4;167(3):124-7. doi: 10.5694/j.1326-5377.1997.tb138809.x. PMID 9269265
- [Background] Butler CC, Rollnick S, Pill R, Maggs-Rapport F, Stott N. Understanding the culture of prescribing: qualitative study of general practitioners' and patients' perceptions of antibiotics for sore throats. BMJ. 1998 Sep 5;317(7159):637-42. doi: 10.1136/bmj.317.7159.637. PMID 9727992
- [Background] Annual report of the chief medical officer, volume two, 2011. Infections and the rise of antimicrobial resistance.
- [Background] WHO Library Cataloguing-in-Publication Data. Antibiotic resistance: Multi-country public awareness survey .World Health Organization. 2015.
- [Background] Lewis MA. Why we must reduce dental prescription of antibiotics: European Union Antibiotic Awareness Day. Br Dent J. 2008 Nov 22;205(10):537-8. doi: 10.1038/sj.bdj.2008.984. PMID 19023306
- [Background] Wise R, Hart T, Cars O, Streulens M, Helmuth R, Huovinen P, Sprenger M. Antimicrobial resistance. Is a major threat to public health. BMJ. 1998 Sep 5;317(7159):609-10. doi: 10.1136/bmj.317.7159.609. No abstract available. PMID 9727981
- [Background] Aljadhey H, Assiri GA, Mahmoud MA, Al-Aqeel S, Murray M. Self-medication in Central Saudi Arabia. Community pharmacy consumers' perspectives. Saudi Med J. 2015 Mar;36(3):328-34. doi: 10.15537/smj.2015.3.10523. PMID 25737176
- [Background] Khan A K A, Banu G, K K R. Antibiotic Resistance and Usage-A Survey on the Knowledge, Attitude, Perceptions and Practices among the Medical Students of a Southern Indian Teaching Hospital. J Clin Diagn Res. 2013 Aug;7(8):1613-6. doi: 10.7860/JCDR/2013/6290.3230. Epub 2013 Jul 1. PMID 24086854
- [Background] Chen C, Chen YM, Hwang KL, Lin SJ, Yang CC, Tsay RW, Liu CE, Young TG. Behavior, attitudes and knowledge about antibiotic usage among residents of Changhua, Taiwan. J Microbiol Immunol Infect. 2005 Feb;38(1):53-9. PMID 15692628
- [Background] Srinivasan A, Song X, Richards A, Sinkowitz-Cochran R, Cardo D, Rand C. A survey of knowledge, attitudes, and beliefs of house staff physicians from various specialties concerning antimicrobial use and resistance. Arch Intern Med. 2004 Jul 12;164(13):1451-6. doi: 10.1001/archinte.164.13.1451. PMID 15249355
- [Background] Vanden Eng J, Marcus R, Hadler JL, Imhoff B, Vugia DJ, Cieslak PR, Zell E, Deneen V, McCombs KG, Zansky SM, Hawkins MA, Besser RE. Consumer attitudes and use of antibiotics. Emerg Infect Dis. 2003 Sep;9(9):1128-35. doi: 10.3201/eid0909.020591. PMID 14519251
- [Background] Azevedo MM, Pinheiro C, Yaphe J, Baltazar F. Portuguese students' knowledge of antibiotics: a cross-sectional study of secondary school and university students in Braga. BMC Public Health. 2009 Sep 23;9:359. doi: 10.1186/1471-2458-9-359. PMID 19775451
- [Background] Simpson SA, Wood F, Butler CC. General practitioners' perceptions of antimicrobial resistance: a qualitative study. J Antimicrob Chemother. 2007 Feb;59(2):292-6. doi: 10.1093/jac/dkl467. Epub 2006 Nov 16. PMID 17110392
- [Background] Wright EP, Jain P. Survey of antibiotic knowledge amongst final year medical students. J Antimicrob Chemother. 2004 Mar;53(3):550-1. doi: 10.1093/jac/dkh096. Epub 2004 Feb 4. No abstract available. PMID 14762052
- [Background] Andre M, Vernby A, Berg J, Lundborg CS. A survey of public knowledge and awareness related to antibiotic use and resistance in Sweden. J Antimicrob Chemother. 2010 Jun;65(6):1292-6. doi: 10.1093/jac/dkq104. Epub 2010 Apr 1. PMID 20360063
- [Background] Armitage, P., Berry, G., & Matthews, J. N. S. Statistical methods in medical research. Wiley Online Library,4rth edition, 2008
- [Result] Mahajan, Dr. Manali. (2014). A Questionnaire based Survey on the Knowledge, Attitude and Practises about Antimicrobial Resistance and Usage among the Second year MBBS Students of a Teaching tertiary care Hospital in Central India. International Journal of Pharmacological Research.